CLINICAL TRIAL: NCT05211518
Title: Preventing IBD Onset in Individuals at Risk
Brief Title: Prevention of Inflammatory Bowel Diseases in Persons at Risk The PIONIR (Preventing IBD Onset in Individuals at Risk) Trial
Acronym: PIONIR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other); The Hospital for Sick Children (Other); The Governors of the University of Alberta (Unknown); University of Manitoba (Other); IWK Health Centre (Other); University of British Columbia (Other); University of Calgary (Other); McGill University (Other); Beilinson Hospital, Petach Tikva,Israel (Unknown)
Responsible Party: Principal Investigator, Dr Dan Turner, Head of The Juliet Keidan Institute of Pediatric Gastroenterology & Nutrition, Shaare Zedek Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PIONIR trial
Record Dates: First submitted 2021-10-04; First posted 2022-01-27 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Chron
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tasty&Healthy (Other): Tasty&Healthy intervention: subjects will receive dietary advice to exclude pro-inflammatory dietary components
  Interventions: Other: Tasty&Healthy
- Habitual diet (Other): Habitual diet: subjects will continue their habitual diet.
  Interventions: Other: Habitual diet

INTERVENTIONS:
Other: Tasty&Healthy — exclude pro-inflammatory dietary components
  Arms: Tasty&Healthy
Other: Habitual diet — subjects will continue their habitual diet.
  Arms: Habitual diet

SUMMARY:
The goal of this study is to explore in a cross over randomized controlled trial, the ability of the Tasty&Healthy dietary intervention (NCT04239248) to alter the parameters associated with future risk of developing Chron's disease (CD) using First Degree Relatives of patients with Crohn's disease, including subjects identified in the Genetic Environmental Microbiome (GEM) Study as having a high-risk score. Specifically, the investigators aim to determine if the Tasty&Healthy dietary intervention can decrease the overall GEM Risk Score (GRS) and/or to alter the individual biological parameters that contribute to this score. The investigators hypothesize that the Tasty&Healthy dietary approach will alter the risk of CD as reflected by a decrease in the GRS.

DETAILED DESCRIPTION:
Several important factors associated with CD onset have already been identified in the GEM analyses, such as elevated faecal calprotectin(FC),altered gut permeability, proteomics, anti-microbial serology, and microbiome composition. These parameters are combined into the GEM Risk Score (GRS).

The first-line therapy in children with CD, according to ECCO/ESPGHAN guidelines, is exclusive enteral nutrition (EEN), meaning 8-12 weeks of exclusive liquid formula. Nutritional therapy may alter intestinal inflammation by several mechanisms, including modulation of the microbiome and an effect on intestinal permeability, both factors assessed in the GEM cohort. EEN is safe and effective, but it is challenging to implement.

Several diets, based on solid foods, have been proposed as alternatives to EEN in an attempt to increase feasibility, three of which have the most data.

Specific carbohydrate diet (SCD) restricts carbohydrates and processed foods and has been long used with variable reported effectiveness.

The CD-TREAT diet induced a positive change to the microbiome, children with active CD entered clinical remission with decreased inflammatory markers.

Crohn's Disease Exclusion Diet (CDED) is based on the exclusion of processed and pro-inflammatory foods, similar to Tasty&Healthy. A recent RCT of CDED diet with 50% liquid formula showed comparable effectiveness as EEN, including normalization of FC and positive effect on the microbiome.

However, the allowed dietary components are not liberal, and the diet is rigid, making it unsuitable as a prevention measure.

In 2014, a cook-book named "Tasty&Healthy" was published as a simple approach to dietary treatment based on the best available evidence. A steering committee of physicians experienced in IBD and nutrition, as well as leading IBD dieticians, reviewed results of dietary studies from animal models, humans and epidemiological cohorts. This review resulted in agreed-upon foods that may aggravate inflammation and thus should be excluded, including all processed and industrialized food, animal fat (dairy, meat), gluten and sugar. Overall, allowed foods in liberal quantities are those prepared at home from readily available ingredients such as fruits, vegetables, fish and shellfish, poultry, oats, eggs, non-gluten grains and legumes. Tasty&Healthy is not a specific diet; it is a dietary approach in which the allowed foods are not structured or restricted. This approach allows flexibility to increase adherence In this study, The Investigators hypothesize that the Tasty&Healthy dietary approach will alter the risk of CD as reflected by a decrease in the GEM CD risk score or alteration of its individual components.

ELIGIBILITY:
Inclusion criteria

* Clinically healthy subjects (i.e. lack of symptoms that may suggest IBD) who are First degree relatives of someone with CD with a high faecal calprotectin (FC)>70μg/g or subjects who have a risk factor for example elevated GRS. Where available LMR will also be assessed to identify subjects ranked as top 100 at risk of CD.
* Younger than 39 years of age, in order to maximize future risk of developing CD.
* No overt ulcerations (other than aphthous ulcerations) in the ileum or colon. Some degree of inflammation may be seen in these high-risk subjects with increased risk parameters and this does not necessarily prompt the diagnosis of CD. Moreover, in this proof of concept study we would like to have those with the highest risk (hence some degree of initial inflammation) but without macroscopic inflammation that clearly is associated with the diagnosis of CD. Patency capsule and VCE procedure will be performed if the subjects calprotectin levels are >70μg/g.

Exclusion Criteria:

* Ulcerative colitis (UC) or IBD-unclassified (IBDU) diagnosis
* The use of antibiotics in the preceding month
* Prior intestinal resection
* Pregnancy (and up until six months after giving birth)
* Celiac disease or Diabetes
* Weight loss or weight gain by more than 20% body weight in the last 3 months
* Extraintestinal manifestations (Arthritis/arthralgia, iritis/uveitis, skin/mouth lesions, peri-anal disease, Other fistula).
* Underweight (children <3th BMI percentile, adult above the age of 18 years: BMI<18.5 kg/m2).

Ages: 6 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The likelihood to develop CD measured by the GRS scale. | 8 weeks of Tasty&Healthy diet.
  Several important factors associated with CD onset have already been identified in the GEM analyses, such as elevated fecal calprotectin (FC), altered gut permeability, proteomics, anti-microbial serology, and microbiome composition. These parameters are potentially modifiable and will be combined into a model to construct the GEM Risk Score (GRS). The range of the GRS is 60.54682691 or higher. The higher the GRS score there is an increased chance of developing Chron's dis.

SECONDARY OUTCOMES:
FC decreased by >30% at the end of the "Tasty&Healthy" intervention, compared to the FC before the intervention. | 8 weeks of Tasty&Healthy diet.
  Decreased level of fecal calprotectin with at least 30% decline from baseline. fecal calprotectin is a test used to detect inflammation in the gastrointestinal tract and is associated with Crohn's disease onset.
Microbiome risk score (MRS) Change in one standard deviation. | 8 weeks of Tasty&Healthy diet.
  Decreased level of Microbiome risk score with at least one standard deviation decline from baseline. The Microbiome risk score is a test we develop to classify individuals according to their risk to develop Crohn's disease onset.
Lactulose-Mannitol Ratio (LMR) Change in one standard deviation. | 8 weeks of Tasty&Healthy diet.
  Decreased level of urinary fractional excretion ratio of Lactulose to Mannitol (LMR) with at least one standard deviation decline from baseline. The LMR is an in vivo test that allow quantification of intestinal barrier permeability that is associated with risk to develop Crohn's disease.
Change in Serum Metabolomics pre and post-intervention | 8 weeks of Tasty&Healthy diet.
  Change in levels of stool, urine, and serum metabolites with at least one standard deviation difference from baseline. Metabolomics allow assessment of host chemical processes involving metabolites, small molecule substrates, intermediates and products of cell or microbial metabolism. Unit of measure is raw area count rescaled to set the median equal to 1.
Change in Serum Proteomics pre and post-intervention | 8 weeks of Tasty&Healthy diet.
  Change in serum proteomics with at least one standard deviation different from baseline. Proteomics allows to assess initiators of most biological processes such as enzymes, cytokines, and transcription factors that contribute to Crohn's disease onset. Unit of measure is normalized protein expression.
Change in Serology pre and post-intervention | 8 weeks of Tasty&Healthy diet.
  Change in antimicrobial antibodies response with at least one standard deviation different from baseline. Serum antimicrobial antibodies allows to assess the immune response against commensal bacteria that are associated with risk of Crohn's disease onset. Unit of measure is titer.
Ability to maintain a balanced diet as measured by food diaries. | 8 weeks of Tasty&Healthy diet.
  Will be assessed by daily caloric intake and nutritional components.
Adherence with the interventions, including assessment of faecal gluten. | 8 weeks of Tasty&Healthy diet.
  Will be assessed using ELISA kit- Buhlman fCAL Elisa
Satisfaction with the treatment received, as assessed by the Satisfaction with Food-Related Life (SFRL) questionnaire. | 8 weeks of Tasty&Healthy diet.
  Will be assessed by the SFRL questionnaire - Grunert KG, Dean M, Raats MM, Nielsen NA, Lumbers M; Food in Later Life Team. A measure of satisfaction with food-related life. Appetite. 2007 Sep;49(2):486-93. doi: 10.1016/j.appet.2007.03.010. Epub 2007 Mar 24. PMID: 17481776.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Turner, Prof, Principal Investigator — Saare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stulman MY, Asayag N, Focht G, Brufman I, Cahan A, Ledderman N, Matz E, Chowers Y, Eliakim R, Ben-Horin S, Odes S, Dotan I, Balicer RD, Benchimol EI, Turner D. Epidemiology of Inflammatory Bowel Diseases in Israel: A Nationwide Epi-Israeli IBD Research Nucleus Study. Inflamm Bowel Dis. 2021 Oct 20;27(11):1784-1794. doi: 10.1093/ibd/izaa341. PMID 33438721
- [Background] Department of Error. Lancet. 2020 Oct 3;396(10256):e56. doi: 10.1016/S0140-6736(20)32028-6. No abstract available. PMID 33010847
- [Background] Beard JA, Franco DL, Click BH. The Burden of Cost in Inflammatory Bowel Disease: A Medical Economic Perspective and the Future of Value-Based Care. Curr Gastroenterol Rep. 2020 Jan 30;22(2):6. doi: 10.1007/s11894-020-0744-z. PMID 32002671
- [Background] Barnes C, Ashton JJ, Borca F, Cullen M, Walker DM, Beattie RM. Children and young people with inflammatory bowel disease attend less school than their healthy peers. Arch Dis Child. 2020 Jul;105(7):671-676. doi: 10.1136/archdischild-2019-317765. Epub 2020 Jan 14. PMID 31937567